CLINICAL TRIAL: NCT01858766
Title: A Phase 2, Multicenter, Randomized, Open-Label Study to Investigate the Safety and Efficacy of Sofosbuvir + GS-5816 for 12 Weeks in Treatment-Naive Subjects With Chronic HCV Infection
Brief Title: Safety and Efficacy of Sofosbuvir + Velpatasvir With or Without Ribavirin in Treatment-Naive Adults With Chronic HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-0102
Record Dates: First submitted 2013-05-10; First posted 2013-05-21 (Estimated); Results first posted 2016-09-15 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2016-07

CONDITIONS: Hepatitis C
Keywords: Hepatitis; HCV Genotype 1; HCV Genotype 2; HCV Genotype 3; HCV Genotype 4; HCV Genotype 5; HCV Genotype 6; treatment naive
MeSH Terms: conditions — Hepatitis C; Hepatitis | interventions — Sofosbuvir; velpatasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (14):
- SOF+VEL 25 mg 12 Weeks (GT1) (Experimental): Participants with genotype 1 HCV infection will receive SOF+VEL 25 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 100 mg 12 Weeks (GT1) (Experimental): Participants with genotype 1 HCV infection will receive SOF+VEL 100 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 25 mg 12 Weeks (GT2/4/5/6) (Experimental): Participants with genotype 2, 4, 5, or 6 HCV infection will receive SOF+VEL 25 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 100 mg 12 Weeks (GT2/4/5/6) (Experimental): Participants with genotype 2, 4, 5, or 6 HCV infection will receive SOF+VEL 100 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 25 mg 12 Weeks (GT3) (Experimental): Participants with genotype 3 HCV infection will receive SOF+VEL 25 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 100 mg 12 Weeks (GT3) (Experimental): Participants with genotype 3 HCV infection will receive SOF+VEL 100 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 25 mg 8 Weeks (GT1) (Experimental): Participants with genotype 1 HCV infection will receive SOF+VEL 25 mg for 8 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 25 mg + RBV 8 Weeks (GT1) (Experimental): Participants with genotype 1 HCV infection will receive SOF+VEL 25 mg plus RBV for 8 weeks.
  Interventions: Drug: SOF; Drug: VEL; Drug: RBV
- SOF+VEL 100 mg 8 Weeks (GT1) (Experimental): Participants with genotype 1 HCV infection will receive SOF+VEL 100 mg for 8 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 100 mg + RBV 8 Weeks (GT1) (Experimental): Participants with genotype 1 HCV infection will receive SOF+VEL 100 mg plus RBV for 8 weeks.
  Interventions: Drug: SOF; Drug: VEL; Drug: RBV
- SOF+VEL 25 mg 8 Weeks (GT2) (Experimental): Participants with genotype 2 HCV infection will receive SOF+VEL 25 mg for 8 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 25 mg + RBV 8 Weeks (GT2) (Experimental): Participants with genotype 2 HCV infection will receive SOF+VEL 25 mg plus RBV for 8 weeks.
  Interventions: Drug: SOF; Drug: VEL; Drug: RBV
- SOF+VEL 100 mg 8 Weeks (GT2) (Experimental): Participants with genotype 2 HCV infection will receive SOF+VEL 100 mg for 8 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 100 mg + RBV 8 Weeks (GT2) (Experimental): Participants with genotype 2 HCV infection will receive SOF+VEL 100 mg plus RBV for 8 weeks.
  Interventions: Drug: SOF; Drug: VEL; Drug: RBV

INTERVENTIONS:
Drug: SOF — 400 mg tablet administered orally once daily
  Other Names: GS-7977; PSI-7977; Sovaldi®
Drug: VEL — Tablet administered orally once daily
  Other Names: GS-5816
Drug: RBV — 200 mg tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Other Names: Ribasphere®
  Arms: SOF+VEL 100 mg + RBV 8 Weeks (GT1); SOF+VEL 100 mg + RBV 8 Weeks (GT2); SOF+VEL 25 mg + RBV 8 Weeks (GT1); SOF+VEL 25 mg + RBV 8 Weeks (GT2)

SUMMARY:
The primary objectives of this study are to evaluate the antiviral efficacy, safety, and tolerability of sofosbuvir (SOF) + velpatasvir (VEL; GS-5816) with or without ribavirin (RBV) in treatment-naive adults with chronic genotype (GT) 1, 2, 3, 4, 5, or 6 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection
* Body mass index (BMI) ≥ 18 kg/m^2
* HCV RNA ≥ 10000 IU/mL at screening
* Use of highly effective contraception methods if female of childbearing potential or sexually active male
* Must not have cirrhosis

Exclusion Criteria:

* Current or prior history of clinically significant illness other than HCV
* Screening ECG with clinically significant abnormalities
* Prior exposure to HCV specific direct acting antiviral agent
* Prior treatment of HCV with interferon or ribavirin
* Pregnant or nursing female or male with pregnant female partner
* Chronic liver disease of non-HCV etiology
* Hepatitis B
* Active drug abuse
* Use of any prohibited concomitant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McNally, PhD, Study Director — Gilead Sciences
Locations (51):
- United States (50):
  - UCSD, La Jolla, California
  - University of California San Diego Medical Center, La Jolla, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Los Angeles Medical Center, Los Angeles, California
  - Ruane Peter J MD Incorporated, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Huntington Medical Research Institutes Liver Center, Pasadena, California
  - Kaiser Permanente Medical Grp, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Kaiser Permante, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Florida Center for Clinical Trials Research, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - South Florida Center of Gastroenterology, P.A, Wellington, Florida
  - Center For Hepatitis C/Atlanta Medical Center, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Indianapolis Gastroenterology & Hepatology, Inc.- ARC, Indianapolis, Indiana
  - Mercy Medical Ctr, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - ID Care, Hillsborough, New Jersey
  - Southwest C.A.R.E. Center, Santa Fe, New Mexico
  - North Shore/Long Island Jewish PRIME, Lake Success, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - UPMC Center For Liver Diseases, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Gastro One, Germantown, Tennessee
  - Nashville Gastrointestinal Specialists Inc., Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Methodist Transplant Physicians, Dallas, Texas
  - Alamo Medical Research, LTD d/b/a American Research Corporation, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - INOVA Institute of Research & Education, Falls Church, Virginia
  - The Liver Institute of Virginia, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Ltd., Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Everson GT, Tran TT, Towner WJ , Davis MN, Wyles D, Nahass R, McNally J, Brainard DM, Han L, Doehle B, Mogalian E, Symonds WT, McHutchison JG, Morgan T, Chung RT. Safety and Efficacy of Treatment with the Interferon-Free, Ribavirin-Free Combination of Sofosbuvir + GS-5816 for 12 Weeks in Treatment Naive Patients with Genotype 1-6 HCV Infection. Journal of Hepatology, Volume 60, Issue 1, Supplement, Page S46. April 2014 (EASL 2014).
- [Result] Tran TT, Morgan TR, Thuluvath PJ, Etzkorn K, Hinestrosa F, Tong M, McNally J, Brainard DM, Han L, Doehle B, Mogalian E, McHutchison JG, Chung RT, Everson GT. Safety and Efficacy of Treatment with Sofosbuvir+ GS-5816±Ribavirin for 8 or 12 Weeks in Treatment Naïve Patients with Genotype 1-6 HCV Infection. Hepatology (2014), 60: 4 (suppl) 237A.
- [Result] Doehle B, Gontcharova V, Chodavarapu1 RK, McNally J, Chung RT, Everson GT, McHutchison JG, Miller MD, Mo H. Resistance Analysis of Treatment-Naive HCV Genotype 1-6 Infected Patients Treated with Sofosbuvir in Combination with GS-5816 for 12 Weeks. Hepatology (2014), 60: 4 (suppl) 1138A.
- [Result] Everson GT, Towner WJ, Davis MN, Wyles DL, Nahass RG, Thuluvath PJ, Etzkorn K, Hinestrosa F, Tong M, Rabinovitz M, McNally J, Brainard DM, Han L, Doehle B, McHutchison JG, Morgan T, Chung RT, Tran TT. Sofosbuvir With Velpatasvir in Treatment-Naive Noncirrhotic Patients With Genotype 1 to 6 Hepatitis C Virus Infection: A Randomized Trial. Ann Intern Med. 2015 Dec 1;163(11):818-26. doi: 10.7326/M15-1000. Epub 2015 Nov 10. PMID 26551051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 22 April 2013. The last study visit occurred on 12 August 2014.
Pre-assignment Details: 469 participants were screened.
Groups:
- SOF+VEL 25 mg 12 Weeks (GT1): Sofosbuvir (SOF) 400 mg tablet + velpatasvir (VEL) 25 mg tablet administered orally once daily for 12 weeks (genotype (GT) 1)
- SOF+VEL 100 mg 12 Weeks (GT1): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 12 weeks (genotype 1)
- SOF+VEL 25 mg 12 Weeks (GT2): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotype 2)
- SOF+VEL 100 mg 12 Weeks (GT2): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 12 weeks (genotype 2)
- SOF+VEL 25 mg 12 Weeks (GT3): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotype 3)
- SOF+VEL 100 mg 12 Weeks (GT3): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 12 weeks (genotype 3)
- SOF+VEL 25 mg 12 Weeks (GT4): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotype 4)
- SOF+VEL 100 mg 12 Weeks (GT4): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 12 weeks (genotype 4)
- SOF+VEL 25 mg 12 Weeks (GT5): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotype 5)
- SOF+VEL 25 mg 12 Weeks (GT6): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotype 6)
- SOF+VEL 100 mg 12 Weeks (GT6): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 12 weeks (genotype 6)
- SOF+VEL 25 mg 8 Weeks (GT1): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 8 weeks (genotype 1)
- SOF+VEL 25 mg + RBV 8 Weeks (GT1): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 8 weeks (genotype 1)
- SOF+VEL 100 mg 8 Weeks (GT1): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 8 weeks (genotype 1)
- SOF+VEL 100 mg + RBV 8 Weeks (GT1): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 8 weeks (genotype 1)
- SOF+VEL 25 mg 8 Weeks (GT2): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 8 weeks (genotype 2)
- SOF+VEL 25 mg + RBV 8 Weeks (GT2): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 8 weeks (genotype 2)
- SOF+VEL 100 mg 8 Weeks (GT2): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 8 weeks (genotype 2)
- SOF+VEL 100 mg + RBV 8 Weeks (GT2): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 8 weeks (genotype 2)
Period: Overall Study
Arm/Group | SOF+VEL 25 mg 12 Weeks (GT1) | SOF+VEL 100 mg 12 Weeks (GT1) | SOF+VEL 25 mg 12 Weeks (GT2) | SOF+VEL 100 mg 12 Weeks (GT2) | SOF+VEL 25 mg 12 Weeks (GT3) | SOF+VEL 100 mg 12 Weeks (GT3) | SOF+VEL 25 mg 12 Weeks (GT4) | SOF+VEL 100 mg 12 Weeks (GT4) | SOF+VEL 25 mg 12 Weeks (GT5) | SOF+VEL 25 mg 12 Weeks (GT6) | SOF+VEL 100 mg 12 Weeks (GT6) | SOF+VEL 25 mg 8 Weeks (GT1) | SOF+VEL 25 mg + RBV 8 Weeks (GT1) | SOF+VEL 100 mg 8 Weeks (GT1) | SOF+VEL 100 mg + RBV 8 Weeks (GT1) | SOF+VEL 25 mg 8 Weeks (GT2) | SOF+VEL 25 mg + RBV 8 Weeks (GT2) | SOF+VEL 100 mg 8 Weeks (GT2) | SOF+VEL 100 mg + RBV 8 Weeks (GT2)
Started | 27 | 28 | 11 | 10 | 27 | 28 | 7 | 7 | 1 | 4 | 5 | 30 | 30 | 29 | 31 | 26 | 25 | 27 | 26
Completed | 26 | 28 | 10 | 10 | 26 | 24 | 7 | 5 | 1 | 4 | 5 | 25 | 25 | 26 | 23 | 20 | 22 | 23 | 22
Not Completed | 1 | 0 | 1 | 0 | 1 | 4 | 0 | 2 | 0 | 0 | 0 | 5 | 5 | 3 | 8 | 6 | 3 | 4 | 4
Not completed — Randomized but Never Treated | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 3 | 5 | 5 | 2 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 1
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug.
Groups:
- SOF+VEL 25 mg 12 Weeks (GT1): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotype 1)
- SOF+VEL 25 mg + RBV 8 Weeks (GT1): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 8 weeks (genotype 1)
- Total: Total of all reporting groups
Arm/Group | SOF+VEL 25 mg 12 Weeks (GT1) | SOF+VEL 100 mg 12 Weeks (GT1) | SOF+VEL 25 mg 12 Weeks (GT2) | SOF+VEL 100 mg 12 Weeks (GT2) | SOF+VEL 25 mg 12 Weeks (GT3) | SOF+VEL 100 mg 12 Weeks (GT3) | SOF+VEL 25 mg 12 Weeks (GT4) | SOF+VEL 100 mg 12 Weeks (GT4) | SOF+VEL 25 mg 12 Weeks (GT5) | SOF+VEL 25 mg 12 Weeks (GT6) | SOF+VEL 100 mg 12 Weeks (GT6) | SOF+VEL 25 mg 8 Weeks (GT1) | SOF+VEL 25 mg + RBV 8 Weeks (GT1) | SOF+VEL 100 mg 8 Weeks (GT1) | SOF+VEL 100 mg + RBV 8 Weeks (GT1) | SOF+VEL 25 mg 8 Weeks (GT2) | SOF+VEL 25 mg + RBV 8 Weeks (GT2) | SOF+VEL 100 mg 8 Weeks (GT2) | SOF+VEL 100 mg + RBV 8 Weeks (GT2) | Total
Number analyzed (Participants) | 27 | 28 | 11 | 10 | 27 | 27 | 7 | 7 | 1 | 4 | 5 | 30 | 30 | 29 | 31 | 26 | 25 | 26 | 26 | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (11.4) | 49 (12.2) | 42 (14.6) | 53 (12.6) | 52 (10.8) | 50 (12.7) | 51 (16.1) | 56 (5.5) | 53 (NA) — N/A because there is only 1 participant in this group. | 57 (4.8) | 54 (9.3) | 50 (10.7) | 53 (8.5) | 55 (9.6) | 52 (13.8) | 52 (10.8) | 54 (11.5) | 54 (10.8) | 51 (9.4) | 52 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 5 | 3 | 9 | 10 | 1 | 3 | 0 | 0 | 1 | 14 | 12 | 13 | 15 | 11 | 8 | 14 | 16 | 159
  Male | 14 | 17 | 6 | 7 | 18 | 17 | 6 | 4 | 1 | 4 | 4 | 16 | 18 | 16 | 16 | 15 | 17 | 12 | 10 | 218
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 2 | 1 | 3 | 2 | 7 | 5 | 39
  Not Hispanic or Latino | 23 | 23 | 10 | 10 | 25 | 26 | 7 | 6 | 1 | 4 | 5 | 26 | 29 | 27 | 30 | 23 | 23 | 19 | 21 | 338
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 6
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Black or African American | 4 | 1 | 0 | 0 | 4 | 0 | 2 | 1 | 0 | 0 | 0 | 4 | 3 | 5 | 5 | 2 | 2 | 2 | 0 | 35
  White | 23 | 25 | 11 | 10 | 22 | 26 | 5 | 5 | 1 | 2 | 1 | 26 | 27 | 24 | 24 | 22 | 23 | 24 | 25 | 326
  Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
HCV Genotype [Number; unit: participants]
  Genotype 1a | 22 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 25 | 24 | 25 | 0 | 0 | 0 | 0 | 142
  Genotype 1b | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 6 | 0 | 0 | 0 | 0 | 32
  Genotype 1g | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Genotype 2 | 0 | 0 | 11 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 25 | 26 | 26 | 124
  Genotype 3 | 0 | 0 | 0 | 0 | 27 | 27 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 54
  Genotype 4 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14
  Genotype 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Genotype 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
IL28b Status [Number; unit: participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 8 | 9 | 1 | 2 | 12 | 13 | 2 | 2 | 1 | 1 | 5 | 9 | 10 | 13 | 9 | 9 | 13 | 9 | 7 | 135
    CT | 16 | 17 | 8 | 8 | 13 | 12 | 5 | 2 | 0 | 3 | 0 | 14 | 16 | 13 | 18 | 14 | 9 | 14 | 14 | 196
    TT | 3 | 2 | 2 | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 7 | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 43
    Missing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.4 (0.60) | 6.4 (0.74) | 6.5 (0.74) | 6.7 (0.78) | 6.4 (1.09) | 6.2 (0.74) | 6.2 (0.58) | 5.8 (0.55) | 7.0 (NA) — N/A because there is only 1 participant in this group. | 6.1 (0.89) | 6.7 (0.88) | 6.5 (0.69) | 6.5 (0.63) | 6.3 (0.85) | 6.6 (0.55) | 6.4 (0.87) | 6.6 (0.80) | 6.5 (0.74) | 6.7 (0.57) | 6.5 (0.75)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 4 | 6 | 2 | 1 | 9 | 6 | 2 | 4 | 0 | 1 | 1 | 5 | 5 | 8 | 3 | 6 | 4 | 5 | 2 | 74
  ≥ 800,000 IU/mL | 23 | 22 | 9 | 9 | 18 | 21 | 5 | 3 | 1 | 3 | 4 | 25 | 25 | 21 | 28 | 20 | 21 | 21 | 24 | 303

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants randomized into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF+VEL 25 mg 12 Weeks (GT1) | SOF+VEL 100 mg 12 Weeks (GT1) | SOF+VEL 25 mg 12 Weeks (GT2) | SOF+VEL 100 mg 12 Weeks (GT2) | SOF+VEL 25 mg 12 Weeks (GT3) | SOF+VEL 100 mg 12 Weeks (GT3) | SOF+VEL 25 mg 12 Weeks (GT4) | SOF+VEL 100 mg 12 Weeks (GT4) | SOF+VEL 25 mg 12 Weeks (GT5) | SOF+VEL 25 mg 12 Weeks (GT6) | SOF+VEL 100 mg 12 Weeks (GT6) | SOF+VEL 25 mg 8 Weeks (GT1) | SOF+VEL 25 mg + RBV 8 Weeks (GT1) | SOF+VEL 100 mg 8 Weeks (GT1) | SOF+VEL 100 mg + RBV 8 Weeks (GT1) | SOF+VEL 25 mg 8 Weeks (GT2) | SOF+VEL 25 mg + RBV 8 Weeks (GT2) | SOF+VEL 100 mg 8 Weeks (GT2) | SOF+VEL 100 mg + RBV 8 Weeks (GT2)
Number analyzed (Participants) | 27 | 28 | 11 | 10 | 27 | 27 | 7 | 7 | 1 | 4 | 5 | 30 | 30 | 29 | 31 | 26 | 25 | 26 | 26
percentage of participants | 96.3 [81.0 to 99.9] | 100.0 [87.7 to 100.0] | 90.9 [58.7 to 99.8] | 100.0 [69.2 to 100.0] | 92.6 [75.7 to 99.1] | 92.6 [75.7 to 99.1] | 100.0 [59.0 to 100.0] | 85.7 [42.1 to 99.6] | 100.0 [2.5 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [47.8 to 100.0] | 86.7 [69.3 to 96.2] | 83.3 [65.3 to 94.4] | 89.7 [72.6 to 97.8] | 80.6 [62.5 to 92.5] | 76.9 [56.4 to 91.0] | 88.0 [68.8 to 97.5] | 88.5 [69.8 to 97.6] | 88.5 [69.8 to 97.6]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- SOF+VEL 25 mg 12 Weeks: SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (all genotypes)
- SOF+VEL 100 mg 12 Weeks: SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 12 weeks (all genotypes)
- SOF+VEL 25 mg 8 Weeks: SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 8 weeks (all genotypes)
- SOF+VEL 25 mg + RBV 8 Weeks: SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 8 weeks (all genotypes)
- SOF+VEL 100 mg 8 Weeks: SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 8 weeks (all genotypes)
- SOF+VEL 100 mg + RBV 8 Weeks: SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 8 weeks (all genotypes)
Arm/Group | SOF+VEL 25 mg 12 Weeks | SOF+VEL 100 mg 12 Weeks | SOF+VEL 25 mg 8 Weeks | SOF+VEL 25 mg + RBV 8 Weeks | SOF+VEL 100 mg 8 Weeks | SOF+VEL 100 mg + RBV 8 Weeks
Number analyzed (Participants) | 77 | 77 | 56 | 55 | 55 | 57
percentage of participants | 0 | 0 | 1.8 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF+VEL 25 mg 12 Weeks (GT1) | SOF+VEL 100 mg 12 Weeks (GT1) | SOF+VEL 25 mg 12 Weeks (GT2) | SOF+VEL 100 mg 12 Weeks (GT2) | SOF+VEL 25 mg 12 Weeks (GT3) | SOF+VEL 100 mg 12 Weeks (GT3) | SOF+VEL 25 mg 12 Weeks (GT4) | SOF+VEL 100 mg 12 Weeks (GT4) | SOF+VEL 25 mg 12 Weeks (GT5) | SOF+VEL 25 mg 12 Weeks (GT6) | SOF+VEL 100 mg 12 Weeks (GT6) | SOF+VEL 25 mg 8 Weeks (GT1) | SOF+VEL 25 mg + RBV 8 Weeks (GT1) | SOF+VEL 100 mg 8 Weeks (GT1) | SOF+VEL 100 mg + RBV 8 Weeks (GT1) | SOF+VEL 25 mg 8 Weeks (GT2) | SOF+VEL 25 mg + RBV 8 Weeks (GT2) | SOF+VEL 100 mg 8 Weeks (GT2) | SOF+VEL 100 mg + RBV 8 Weeks (GT2)
Number analyzed (Participants) | 27 | 28 | 11 | 10 | 27 | 27 | 7 | 7 | 1 | 4 | 5 | 30 | 30 | 29 | 31 | 26 | 25 | 26 | 26
percentage of participants
  SVR4 | 96.3 [81.0 to 99.9] | 100.0 [87.7 to 100.0] | 90.9 [58.7 to 99.8] | 100.0 [69.2 to 100.0] | 92.6 [75.7 to 99.1] | 100.0 [87.2 to 100.0] | 100.0 [59.0 to 100.0] | 85.7 [42.1 to 99.6] | 100.0 [2.5 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [47.8 to 100.0] | 86.7 [69.3 to 96.2] | 83.3 [65.3 to 94.4] | 93.1 [77.2 to 99.2] | 87.1 [70.2 to 96.4] | 88.5 [69.8 to 97.6] | 88.0 [68.8 to 97.5] | 92.3 [74.9 to 99.1] | 88.5 [69.8 to 97.6]
  SVR24 | 92.6 [75.7 to 99.1] | 100.0 [87.7 to 100.0] | 90.9 [58.7 to 99.8] | 100.0 [69.2 to 100.0] | 92.6 [75.7 to 99.1] | 92.6 [75.7 to 99.1] | 100.0 [59.0 to 100.0] | 85.7 [42.1 to 99.6] | 100.0 [2.5 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [47.8 to 100.0] | 86.7 [69.3 to 96.2] | 83.3 [65.3 to 94.4] | 89.7 [72.6 to 97.8] | 80.6 [62.5 to 92.5] | 76.9 [56.4 to 91.0] | 88.0 [68.8 to 97.5] | 88.5 [69.8 to 97.6] | 88.5 [69.8 to 97.6]

4. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+VEL 25 mg 12 Weeks (GT1) | SOF+VEL 100 mg 12 Weeks (GT1) | SOF+VEL 25 mg 12 Weeks (GT2) | SOF+VEL 100 mg 12 Weeks (GT2) | SOF+VEL 25 mg 12 Weeks (GT3) | SOF+VEL 100 mg 12 Weeks (GT3) | SOF+VEL 25 mg 12 Weeks (GT4) | SOF+VEL 100 mg 12 Weeks (GT4) | SOF+VEL 25 mg 12 Weeks (GT5) | SOF+VEL 25 mg 12 Weeks (GT6) | SOF+VEL 100 mg 12 Weeks (GT6) | SOF+VEL 25 mg 8 Weeks (GT1) | SOF+VEL 25 mg + RBV 8 Weeks (GT1) | SOF+VEL 100 mg 8 Weeks (GT1) | SOF+VEL 100 mg + RBV 8 Weeks (GT1) | SOF+VEL 25 mg 8 Weeks (GT2) | SOF+VEL 25 mg + RBV 8 Weeks (GT2) | SOF+VEL 100 mg 8 Weeks (GT2) | SOF+VEL 100 mg + RBV 8 Weeks (GT2)
Number analyzed (Participants) | 27 | 28 | 11 | 10 | 27 | 27 | 7 | 7 | 1 | 4 | 5 | 30 | 30 | 29 | 31 | 26 | 25 | 26 | 26
percentage of participants | 3.7 | 0 | 0 | 0 | 7.4 | 7.4 | 0 | 0 | 0 | 0 | 0 | 10.0 | 16.7 | 10.3 | 16.1 | 23.1 | 8.0 | 11.5 | 11.5

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF+VEL 25 mg 12 Weeks | SOF+VEL 100 mg 12 Weeks | SOF+VEL 25 mg 8 Weeks | SOF+VEL 25 mg + RBV 8 Weeks | SOF+VEL 100 mg 8 Weeks | SOF+VEL 100 mg + RBV 8 Weeks
Serious Adverse Events (participants affected / at risk) | 2/77 | 1/77 | 3/56 | 1/55 | 0/55 | 0/57
Other Adverse Events (participants affected / at risk) | 38/77 | 45/77 | 27/56 | 43/55 | 22/55 | 36/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+VEL 25 mg 12 Weeks (N=77) | SOF+VEL 100 mg 12 Weeks (N=77) | SOF+VEL 25 mg 8 Weeks (N=56) | SOF+VEL 25 mg + RBV 8 Weeks (N=55) | SOF+VEL 100 mg 8 Weeks (N=55) | SOF+VEL 100 mg + RBV 8 Weeks (N=57)
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+VEL 25 mg 12 Weeks (N=77) | SOF+VEL 100 mg 12 Weeks (N=77) | SOF+VEL 25 mg 8 Weeks (N=56) | SOF+VEL 25 mg + RBV 8 Weeks (N=55) | SOF+VEL 100 mg 8 Weeks (N=55) | SOF+VEL 100 mg + RBV 8 Weeks (N=57)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 4 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 1 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 9 | 6 | 1 | 3 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 7 | 3 | 5 | 2 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 4 | 0 | 4 | 1 | 4
Nausea (Gastrointestinal disorders) | 10 | 8 | 4 | 7 | 7 | 8
Vomiting (Gastrointestinal disorders) | 5 | 1 | 0 | 0 | 0 | 4
Fatigue (General disorders) | 19 | 14 | 7 | 17 | 2 | 21
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 2 | 1 | 3
Nasopharyngitis (Infections and infestations) | 2 | 5 | 6 | 4 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 1 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 2 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 4 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 2 | 2 | 0 | 3
Headache (Nervous system disorders) | 16 | 14 | 7 | 21 | 9 | 10
Anxiety (Psychiatric disorders) | 6 | 1 | 2 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 3 | 3 | 9 | 1 | 5
Irritability (Psychiatric disorders) | 4 | 1 | 1 | 5 | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 4 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 4 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2 | 3 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 2 | 3 | 0 | 5
Rash (Skin and subcutaneous tissue disorders) | 4 | 4 | 1 | 7 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years